CLINICAL TRIAL: NCT01073618
Title: Post Marketing Surveillance Study To Observe The Safety And Efficacy Of Vfend® IV
Brief Title: Non-Interventional Post Marketing Surveillance Study To Observe The Safety And Efficacy Of Vfend® IV
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A1501067
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Results first posted 2010-09-16 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-05

CONDITIONS: Serious Fungal Infections
Keywords: voriconazole; Korea; invasive fungal infection
MeSH Terms: conditions — Invasive Fungal Infections | interventions — Voriconazole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A.: Patients who are indicated for VFEND according to drug package insert.
  Interventions: Drug: voriconazole IV

INTERVENTIONS:
Drug: voriconazole IV — 6 mg/kg iv q 12 hours (loading) then maintenance
  Other Names: Vfend

SUMMARY:
This is non-interventional study of voriconazole IV formulation in clinical use, which was mandated by the Korean government agency following the approval of Vfend in the Republic of Korea.

ELIGIBILITY:
Inclusion Criteria:

* Invasive aspergillosis and other serious fungal infections.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are indicated for VFEND according to drug package insert.
Sampling Method: Non-Probability Sample
Enrollment: 692 (Actual)
Dates: Start 2006-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1501067&StudyName=Non-Interventional%20Post%20Marketing%20Surveillance%20Study%20To%20Evaluate%20The%20Safety%20And%20Efficacy%20Of%20Vfend%AE%20IV

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 692 participants enrolled in this study. Of these, 379 participants were treated with the IV formulation of Vfend only, and 313 participants were treated with Vfend IV and Vfend tablets sequentially or vice versa. These 313 participants are also included in study A1501068 (NCT01073631).
Groups:
- Vfend: Vfend (voriconazole) intravenous (IV) for use as indicated according to the approved local product document (LPD) or sequential IV and Vfend tablets treatment (or vice versa) for use as indicated according to approved LPD.
Period: Overall Study
Arm/Group | Vfend
Started | 692
Completed | 385
Not Completed | 307
Not completed — Death | 208
Not completed — Adverse Event | 19
Not completed — Other | 80

BASELINE CHARACTERISTICS:
Arm/Group | Vfend
Number analyzed (Participants) | 692
Age, Customized [Number; unit: participants]
  <18 years | 97
  Between 18 and 44 years | 218
  Between 45 and 64 years | 282
  >=65 years | 95
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 275
  Male | 417

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Categorical Clinical Response: Cure, Improvement, Failure, or Unevaluable
Description: Clinical response defined as: Cure=resolution of all baseline signs and symptoms of fungal infection(s); Improvement=lessening of baseline signs and symptoms or absence of one or more, but not all baseline findings; Failure=no improvement or deterioration of baseline condition; Unevaluable=incomplete therapy (efficacy could not be evaluated or discontinuation was not followed up).
Time Frame: Baseline (Day 1) up to 2 years
Population: Safety population: participants received at least 1 dose of study drug for the approved indication (=Intent to treat [ITT] population plus all unevaluable participants); ITT=participants received study drug for the approved indication and had been evaluated for related parameters at least once.
Measure: Number; unit: percentage of participants
Arm/Group | Vfend
Number analyzed (Participants) | 692
percentage of participants
  Cure | 12.72
  Improvement | 41.47
  Failure | 17.92
  Unevaluable | 27.89
Statistical Analysis 1: Comparison: Vfend; Efficacy Rate (treatment effective) = Percentage of evaluable participants with clinical response of cure or improvement; Test type: Superiority or Other; Normal approximation to binomial; Efficacy rate (percent) = 75.15, 95% CI 2-sided [71.36 to 78.94] — Confidence Interval (CI) by normal approximation to binomial

2. Secondary Outcome: Percentage of Participants With Cultivated Strain Mycological Response: Eradication, Persistence, Superinfection, or Not Evaluable
Description: In case cultivation performed, cultivated strain before and after Vfend administration recorded, and the improvement of mycological outcomes after administration evaluated. Mycological response defined as: Eradication=absence of signs and symptoms of fungal infection; Persistence=(no eradication) presence of fungal infection; Superinfection=existence of different strains from strains separated prior to study medication; Not evaluable=a follow-up mycological cultivation is not performed.
Time Frame: Baseline (Day 1) up to 2 years
Population: ITT; N=number of subjects evaluated for mycological response.
Measure: Number; unit: percentage of participants
Arm/Group | Vfend
Number analyzed (Participants) | 159
percentage of participants
  Eradication | 64.78
  Persistence | 27.67
  Superinfection | 3.77
  Not evaluable | 3.77

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events are reported from the time of the first dose of study treatment up to 28 days after last dose of study treatment.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Vfend
Serious Adverse Events (participants affected / at risk) | 239/692
Other Adverse Events (participants affected / at risk) | 94/692
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vfend (N=692)
Anaemia (Blood and lymphatic system disorders) | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Neutropenic colitis (Gastrointestinal disorders) | 1
Brain death (General disorders) | 1
Condition aggravated (General disorders) | 1
Disease progression (General disorders) | 3
General physical health deterioration (General disorders) | 1
Multi-organ failure (General disorders) | 17
Pyrexia (General disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 3
Hepatic function abnormal (Hepatobiliary disorders) | 4
Hepatorenal failure (Hepatobiliary disorders) | 1
Hepatosplenomegaly (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Acute graft versus host disease in intestine (Immune system disorders) | 2
Acute graft versus host disease in skin (Immune system disorders) | 1
Graft versus host disease (Immune system disorders) | 2
Anal abscess (Infections and infestations) | 1
Aspergillosis (Infections and infestations) | 6
Brain abscess (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cytomegalovirus infection (Infections and infestations) | 2
Enterococcal sepsis (Infections and infestations) | 2
Fungal infection (Infections and infestations) | 2
Liver abscess (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 54
Pneumonia fungal (Infections and infestations) | 2
Pneumonia primary atypical (Infections and infestations) | 1
Sepsis (Infections and infestations) | 25
Septic shock (Infections and infestations) | 43
Collapse of lung (Injury, poisoning and procedural complications) | 1
Acoustic stimulation tests (Investigations) | 1
Blood creatinine (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Cytomegalovirus test positive (Investigations) | 2
Liver function test abnormal (Investigations) | 1
Oxygen saturation decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Transaminases increased (Investigations) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 3
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leukaemic infiltration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 2
Cerebral infarction (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 8
Haemorrhage intracranial (Nervous system disorders) | 1
Intracranial pressure increased (Nervous system disorders) | 1
Paraplegia (Nervous system disorders) | 1
Azotaemia (Renal and urinary disorders) | 3
Cystitis haemorrhagic (Renal and urinary disorders) | 1
Nephropathy toxic (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 3
Renal failure acute (Renal and urinary disorders) | 9
Renal failure chronic (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 12
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 9
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 6
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 2
Hypotension (Vascular disorders) | 3
Shock (Vascular disorders) | 1
Euthyroid sick syndrome (Endocrine disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Enterococcal infection (Infections and infestations) | 1
Chemical peritonitis (Injury, poisoning and procedural complications) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mental impairment (Nervous system disorders) | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vfend (N=692)
Diarrhoea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 7
Pyrexia (General disorders) | 12
Hyperbilirubinaemia (Hepatobiliary disorders) | 14
Blood creatinine increased (Investigations) | 10
Liver function test abnormal (Investigations) | 14
Transaminases increased (Investigations) | 10
Hypokalaemia (Metabolism and nutrition disorders) | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 7
Hypertension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.